CLINICAL TRIAL: NCT05276388
Title: Establishment of a Biological Biobank of Subjects Vaccinated Against SARS-Cov-2 Infection (COVID-BioVac)
Brief Title: Establishment of a Biological Biobank of Subjects Vaccinated Against SARS-CoV-2 Infection (COVID-19)
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Ciceri Fabio, Principal Investigator, Professor and Head of Hematology, IRCCS San Raffaele
Other Study IDs: COVID BioVAC
Record Dates: First submitted 2022-03-07; First posted 2022-03-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Coronavirus Infections
Keywords: Biobank; SARS-CoV-2; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: biological bank — biological bank of subjects vaccinated against SARS-CoV-2 infection

SUMMARY:
Establishment of a biological bank of subjects vaccinated against SARS-Cov-2 infection (COVID-BioVac)

DETAILED DESCRIPTION:
The purpose of the COVID-BioVac study is to establish a biobank of biological samples from subjects who have received the anti-SARS-CoV-2 vaccine, with the ultimate aim (following approval by the EC of specific substudies) to study and characterize the antiviral immune response generated following anti-SARS-CoV-2 vaccination. To this end, the COVID-BioVac Biobank will be officially established for the collection and storage of human biological material, non-profit, to support research activities aimed at advancing scientific knowledge, including in the genetic field, on the immune response. vaccination-induced anti-SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Who have vaccinated for SARS-CoV-2 with Pfizer-BioNTech vaccine or others
* Signing of informed consent from January to March 2021

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees, fellows, collaborators of the San Raffaele Hospital and other subjects who will be deemed suitable
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccines response | from Day 1 of first vaccination up to 1 years after the last vaccination
  Create a Biobank to evaluate the immunogenicity of COVID-19 vaccines in terms of antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Rovere Querini, MD, Study Chair — IRCCS Ospedale San Raffaele; Massimo Locatelli, MD, Study Chair — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No